CLINICAL TRIAL: NCT03661125
Title: A Randomised, Balanced, Double-blind Two-way Crossover Design Study to Evaluate the Effects of SRC Kinase Inhibitor, Saracatinib, on Brain Activity Associated With Visual Processing in Patients With Parkinson's Disease Psychosis.
Brief Title: SRC Inhibition as a Potential Target for Parkinson's Disease Psychosis
Acronym: SCRIPT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: AstraZeneca (Industry); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 247303
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease Psychosis
MeSH Terms: interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saracatinib or placebo (Experimental): In the first arm of the study, participants will be randomised into either the group that receives Saracatinib (study drug) or the Placebo.
  Interventions: Drug: Saracatinib; Drug: Placebo Oral Tablet
- Placebo or Saracatinib (Cross-over) (Experimental): The groups will now cross over i.e. the group that had the study drug in the first arm will get the placebo in the second arm and the group that had the placebo in the first arm will have the study drug in the second arm.
  Interventions: Drug: Saracatinib; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Saracatinib — AZD0530 (Saracatinib) 50 mg Tablet Pink Round 7.0 mm ADM P/5406/49. Two tablets to be taken every morning for 14 days.
Drug: Placebo Oral Tablet — Placebo AZD0530 (Saracatinib) 50 mg Tablet Pink Round 7.0 mm ADM P/5406/37. Two tablets to be taken every morning for 14 days.

SUMMARY:
Parkinson's disease is often characterised by movement symptoms such as rigidity and bradykinesia, however, there are a number of non-motor symptoms that can have a significant impact on quality of life. One of the most common non-motor symptoms of Parkinson's disease is visual hallucinations (where someone sees things that don't exist outside their mind). . Recent findings led to the approval of a drug called Pimavanserin as a treatment for PD psychosis in the USA. Based on other recent studies, we believe that Saracatinib, a drug that interacts within the same system as Pimavanserin, is a potential treatment for PD psychosis. Saracatinib has shown to reduce the intensity of the psychedelic effect induced by psilocybin (a naturally occurring psychedelic found in psilocybe mushrooms) and attenuate social cognition and brain changes in healthy volunteers. The aim of this study is to test the effects of 14 days dosing of saracatinib or placebo on 30 volunteers with PD psychosis. We aim to to use neuroimaging combined with psychopharmacology to provide evidence that a putative new treatment approach can modulate abnormal visual cortex activation in patients with PD psychosis. If positive, this proof of mechanism study would provide a strong platform to pursue symptom modification studies with Saracatinib.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative condition which has a 1% prevalence in the over 60s and also affects young adults. As well as motor symptoms such as akinesia or rigidity, many patients also experience non-motor symptoms of which psychosis is the most common (Chang and Fox, 2016). Current treatments for Parkinson's disease psychosis include atypical antipsychotics such as quetiapine, clozapine and pimavanserin (a 5-HT2a inverse agonist). Pimavanserin has recently been approved in the USA as a PD psychosis treatment; it has been shown to have an overall effect on reducing hallucinations as a whole, but not on visual hallucinations specifically. Functional neuroimaging evidence confirms dysfunctional ventral visual pathway activity in PD psychosis with altered metabolism, blood flow and brain activation following visual stimulation (Chang and Fox, 2016). Outside of the ventral visual pathways, two imaging studies in PD patients with visual hallucinations have shown altered connectivity within the default mode network, a brain system implicated in many neuropsychiatric conditions, pointing to more widespread abnormalities (Chang and Fox, 2016). Structural imaging studies show some atrophy within the ventral visual pathways, but also implicates brain regions outside of visual processing areas, including parietal, frontal, and cerebellar and hippocampal regions (Ffytche et al., 2017). Moreover, even though the serotoninergic dysfunction underpinning Parkinson's disease psychosis is not fully understood, animal studies with psychedelics have pointed to the dimerisation of the 5-HT2A and mGlu2 receptors and the over recruitment of specific downstream signalling pathways. Src kinase inhibition is a potential mechanism for blocking the hallucinogenic effects of 5-HT2A receptor agonism. Src kinase inhibitor, Saracatinib, has shown to reduce the intensity of the psychedelic effect induced by psilocybin (a naturally occurring psychedelic found in psilocybe mushrooms (Byock, 2018)) and attenuate social cognition and brain changes in healthy volunteers. We will test the effects of Saracatinib on brain activity associated with visual processing using a visual processing task, known to be sensitive to 5-HT2a receptor stimulation in previous studies with psilocybin (Carter et al., 2004), and a visual recognition task (Meppelink et al., 2009) with known sensitivity to PD psychosis, both scanned using the latest implementation of multi-echo blood oxygen level dependent (BOLD) functional Magnetic Resonance Imaging (fMRI). We aim to conduct a double-blind crossover design study, looking at the effects of Saracatinib and placebo treatment on 26 patients who have PD with psychosis. Existing data shows that 10 days of dosing with Saracatinib will achieve a steady state level that is known to be well tolerated in people with Alzheimer's disease (Nygaard et al., 2015). Therefore, participants will be given an oral dose of 100mg of Saracatinib or placebo as two 50mg tablets to be taken once daily for 14 days. Participants will return to the clinic on day 14 for their final dose of Saracatinib or placebo, fMRI and EEG scans, cognitive assessments, physical examination and blood screen. The participants will then move onto the second treatment arm where they will receive a further 14 days of dosing with saracatinib or placebo depending on the group they were in for the first treatment arm. There will be a minimum 2-week washout between treatment arms to avoid potential carry over effects.

ELIGIBILITY:
Inclusion Criteria:

* Understand the study procedures and agree to participate by providing written informed consent.
* Have a confirmed diagnosis of Parkinson's disease using internationally accepted UK brain bank criteria.
* Be male or female
* Be right handed
* Aged 40 years or over
* Be judged to be in good health by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12 lead ECG and vital signs measurements performed at screening and prior to administration of the initial dose of study drug.
* Have a score of at least 22 on the Montreal Cognitive Assessment (MoCA).
* Have a diagnosis of idiopathic PD with moderate severity
* Have a combined score of at least 6 or an individual score of at least 4 on the neuropsychiatric inventory (NPI [20]) 23 items A (delusions) and/or B (hallucinations).

Exclusion Criteria:

* Is a female of child bearing potential
* Is currently taking anticholinergic medication
* Is currently taking any medication known to be a moderate or potent CYP3A4 inducer or inhibitor.
* Has an ongoing disability, medical or neurological history, cognitive impairment, or conditions that in the opinion of the investigator may interfere with study conduct or clinical assessments.
* Refuses to be withdrawn from quetiapine (see section 4.7).
* Has a family history of psychosis in a first degree relative
* Has poor peripheral arterial/venous access or recent wrist trauma that will restrict ability to gain venous access.
* Is currently using prescription or non-prescription drugs and herbal supplements, which are deemed to affect the integrity of the study, within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication. As an exception, paracetamol or acetaminophen may be used at doses of 1 g/day.
* Has a history of sensitivity to any of the study medications or any of the excipient constituents.
* Has a history of febrile illness within 5 days prior to the first dose
* Has a hairstyle which would affect EEG recording.
* Has any condition possibly affecting drug absorption (eg, gastrectomy).
* Has a history of regular alcohol consumption exceeding 14 units/week (6 glasses of 13.0% wine (175ml), 6 pints of 4.0% lager or ale (568ml), 5 pints of 4.5% cider (568 ml) or 14 glasses of 10.0% spirits (25ml)) within 6 months of screening.
* Uses tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Uses caffeine containing products of the equivalence of 5 cups of regular filter coffee per day
* Has a positive urine drug screen on or after the screening visit during their active involvement in the study for opiates, methadone, cocaine, amphetamines (including MDMA), barbiturates, benzodiazepines and cannabinoids.
* Is unwilling or unable to comply with the Lifestyle guidelines.
* Has, in the opinion of the investigator, has any medical or psychological condition or social circumstances which would impair their ability to participate reliably in the study, or who may increase the risk to themselves or others by participating.
* Is male and is unwilling to follow the contraception guidance or has a female partner of child bearing potential who is unwilling to follow the contraception guidance throughout the study.
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN)
* Total bilirubin > 1.25 x ULN
* Known congenital long QT syndrome
* Baseline resting QTcF > 470ms on 12 lead ECG
* Positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody at screening
* Known to have tested positive for human immunodeficiency virus.
* Participation in another clinical study with an investigational product administered in the last 3 months
* Below the lower limit of normal Hb, total WBC and neutrophils on blood counts as per the reference ranges of the laboratory conducting the tests.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference between study drug and placebo in BOLD activity in the ventral visual stream during visual recognition vs. the control task measure using fMRI | 2 months (two treatment arms)
  Using functional magnetic resonance imaging (fMRI) to look at the effect of saracatinib in attenuating the reduced response in the ventral visual stream on the visual recognition tasks, compared to placebo.

SECONDARY OUTCOMES:
Difference between study drug and placebo in BOLD activity in the occipito-temporal region during the visual processing task (Kanisza illusion) | 2 months (two treatment arms)
  Using functional magnetic resonance imaging (fMRI) to look at the difference in blood oxygen level dependent activity in the occipito-temporal regions between Saracatinib and placebo during a visual processing task that involves looking and making decisions about a visual illusion that involves shapes that create the illusion of edges that do not exist physically
Change in Mismatch negativity (MMN) in microvolts (mV) and connectivity with the posterior cingulate hub of the default mode network | 2 months (two treatment arms)
  Using electroencephalogram (EEG) to look at change in brain activity within specific areas of the brain that are known to work together.

OTHER OUTCOMES:
Seed-based connectivity from the Regions of Interest (ROI) within the inferotemporal cortex. | 2 months (two treatment arms)
  Using fMRI to look at connectivity within the inferotemporal cortex.
Difference between study drug and placebo in MMN amplitude at FZ on EEG. | 2 months (two treatment arms)
Test a prediction error model for the effects of Saracatinib on brain activity during a mismatch negativity paradigm on the EEG. | 2 months (two treatment arms)
Difference between study drug and placebo in Factor summary score on the scales for assessment of positive symptoms in Parkinson's disease (SAPS-PD) and the Neuropsychiatric Inventory (NPI). | 2 months (two treatment arms)
  Scale for the Assessment of Positive Symptoms- Parkinson's Disease (SAPS-PD)- a 9 question scale that asks about the most frequently reported non-motor symptoms of Parkinson's disease including visual hallucinations and delusions and the severity of symptoms.
  Neuropsychiatric Inventory (NPI)- an informant-based scale that was developed to assess neuropsychiatric symptoms. It consists of 12 items, but section A and B are delusions and hallucinations respectively. If symptoms are present, then more information is obtained through questions about frequency (scale of 1-3) and severity (scale of 1-4). The total scores are added up to get the NPI total score.

CONTACTS AND LOCATIONS:
Overall Officials: Mitul Mehta, Principal Investigator — King's College London
Locations (1):
- Mitul Mehta, London, Camberwell, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Our consent procedures include asking for permission to share anonymised data with other researchers. If consent is given then the anonymised data will be added to our database. Currently interested researchers need to apply for accessto our database.

REFERENCES:
- [Background] Nygaard HB, Wagner AF, Bowen GS, Good SP, MacAvoy MG, Strittmatter KA, Kaufman AC, Rosenberg BJ, Sekine-Konno T, Varma P, Chen K, Koleske AJ, Reiman EM, Strittmatter SM, van Dyck CH. A phase Ib multiple ascending dose study of the safety, tolerability, and central nervous system availability of AZD0530 (saracatinib) in Alzheimer's disease. Alzheimers Res Ther. 2015 Apr 14;7(1):35. doi: 10.1186/s13195-015-0119-0. eCollection 2015. PMID 25874001
- [Background] Chang A, Fox SH. Psychosis in Parkinson's Disease: Epidemiology, Pathophysiology, and Management. Drugs. 2016 Jul;76(11):1093-118. doi: 10.1007/s40265-016-0600-5. PMID 27312429
- [Background] Ffytche DH, Creese B, Politis M, Chaudhuri KR, Weintraub D, Ballard C, Aarsland D. The psychosis spectrum in Parkinson disease. Nat Rev Neurol. 2017 Feb;13(2):81-95. doi: 10.1038/nrneurol.2016.200. Epub 2017 Jan 20. PMID 28106066
- [Background] Byock I. Taking Psychedelics Seriously. J Palliat Med. 2018 Apr;21(4):417-421. doi: 10.1089/jpm.2017.0684. Epub 2018 Jan 22. PMID 29356590
- [Background] Carter OL, Pettigrew JD, Burr DC, Alais D, Hasler F, Vollenweider FX. Psilocybin impairs high-level but not low-level motion perception. Neuroreport. 2004 Aug 26;15(12):1947-51. doi: 10.1097/00001756-200408260-00023. PMID 15305143
- [Background] Meppelink AM, de Jong BM, Renken R, Leenders KL, Cornelissen FW, van Laar T. Impaired visual processing preceding image recognition in Parkinson's disease patients with visual hallucinations. Brain. 2009 Nov;132(Pt 11):2980-93. doi: 10.1093/brain/awp223. Epub 2009 Sep 15. PMID 19755518

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT03661125/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT03661125/ICF_001.pdf